CLINICAL TRIAL: NCT01943123
Title: Effect of Commercially Available Probiotic Drink on Number of Salivary Mutans Streptococci in School Going Children Aged 12-14 Years in Bangalore City (India): Randomized Controlled Trial
Brief Title: Effect of Probiotic Drink on Number of Salivary Mutans Streptococci in School Going Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Oxford Dental College, Hospital and Research Center, Bangalore, India (Other)
Responsible Party: Principal Investigator, Dr. Aman deep Pabbla, assistant professor, The Oxford Dental College, Hospital and Research Center, Bangalore, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: vani-1
Record Dates: First submitted 2013-09-05; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Dental Caries
Keywords: probiotics,; streptococcus mutans,; lactobacilli,; plaque index,; gingival index
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotic drink (Experimental): experimental group (30 subjects) were given 50 ml of probiotic drink for 6 months on daily basis
  Interventions: Dietary Supplement: probiotic drink
- plain, unsweetend, unflavored pasturised milk (Placebo Comparator): control group/ placebo group (30 subjects) were given pasteurized milk (50 ml) for 6 months on regular basis
  Interventions: Dietary Supplement: Placebo Comparator: plain, unsweetend, unflavored pasturised milk

INTERVENTIONS:
Dietary Supplement: probiotic drink — comparison of study group (probiotic group) with the control group regarding the number of CFU of microbes in oral cavity and the overall oral health status measured using indices
  Other Names: yakult probiotic drink
  Arms: probiotic drink
Dietary Supplement: Placebo Comparator: plain, unsweetend, unflavored pasturised milk — comparison of control group with the study group (probiotic group) regarding the number of CFU of microbes in oral cavity and the overall oral health status measured using indices
  Arms: plain, unsweetend, unflavored pasturised milk

SUMMARY:
This study was conducted to assess the effects of commercially available probiotic drink on the number of salivary mutans streptococci in school going children, aged 12-14 years in Bangalore city in India

DETAILED DESCRIPTION:
Probiotic bacteria are thought to reduce the risk of diseases in oral cavity, namely dental caries. Studies have suggested that oral cavity can benefit immensely from these friendly bacteria, although more clinical trials are needed to establish concrete results. Hence, this study was undertaken as a 6 month clinical trial to assess the effects of probiotic on the most frequent resident of oral micro flora- the mutans streptococci.

Method- Design: parallel arm design Sample size: 60 subjects (30 subjects in each group) Duration: 6 months

Material used- Intervention/manipulation: 50ml commercially available probiotic drink for one group (30 subjects in study group) and 50 ml of plain, unsweetened and unflavored milk to control group (30 subjects in control group)for a period of 6 months.

Indices used: plaque index- Turskey Gilmore-Glikman modification of Quigley-Hein, Plaque Index (1970)

Gingival Index-Loe.H and Silness P. gingival index (1963)

Both the indices were used twice, at the start of the study, that is, to collect base line data and at the end of the intervention period (6 months)as final data collected.

Sample collection: stimulated saliva was collected (5ml) and analyzed for CFU of streptococcus mutans and lactobacilli at the start of the study and after 6 months, at the end of the intervention.

Statistical analysis: students t test, fisher exact test and chi-square test were used to compare the baseline data with the final data collected at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* no active carious lesion
* restored dental cavities
* on no systemic antibiotic medication 6 weeks before commencing the study

Exclusion Criteria:

* habitual consumers of probiotics or xylitol chewing gums
* recent exposure to topical/ systemic fluoride treatment
* undergoing any orthodontic treatment during the entire study tenure

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
saliva samples were tested for CFU for streptococci mutans and lactobacilli | feburary 2011 and july 2011 (6 months)
  Saliva samples were tested and the results reveled that number of CFU for both streptococci mutans and lactobacilli varied significantly at the baseline and post intervention in study group (subjects who received probiotic drink). There was reduction in number of CFU of streptococci mutans and lactobacilli in study group.

OTHER OUTCOMES:
plaque and gingival indices were used | feburary 2011- july 2011 (6 months)
  Plaque index- Turskey Gilmore-Glikman modification of Quigley-Hein, Plaque Index (1970)and Gingival Index-Loe.H and Silness P. Gingival index (1963)were used at the beginning of the study and after the intervention was over, the indices were again used to collect the final data. Significant reduction in the mean scores was observed for both the indices in study group (the subjects who were given probiotic drink)whereas the results did not vary markedly in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: vani shree nanjundaiah, MDS, Study Director — The Oxford Dental College, Bangalore, India
Locations (1):
- The Oxford Dental College, Bangalore, Karnataka, India